CLINICAL TRIAL: NCT04414709
Title: Evaluation of Short Implants' Success for Teeth Replacement in Atrophic Posterior Mandibular Ridge (A Clinical Trial)
Brief Title: Evaluation of Short Implants' Success for Teeth Replacement in Atrophic Posterior Mandibular Ridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, fady michel tadros hanna, Oral Surgery Master's student, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IORG 0008839
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Alveolar Bone Loss
Keywords: Short implant; Splinted short implant
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two short implants (Experimental): DENTIUM superline implant fixture is characterized by sandblasted with large grits and acid etched surface treatment (S.L.A). SLA surface allows good bone-implant contact with good clinical performance, maintaining crestal bone margin. Short Implants of 7.0 mm length and 4.5 mm diameter are to be used. The Short Implants are characterized by 1.5mm supra-bony smooth collar, and 5.5mm infra-bony surface treated double threaded titanium.
  Interventions: Other: Double short implant
- Single short implant (Active Comparator): DENTIUM superline implant fixture is characterized by sandblasted with large grits and acid etched surface treatment (S.L.A). SLA surface allows good bone-implant contact with good clinical performance, maintaining crestal bone margin. Short Implants of 7.0 mm length and 4.5 mm diameter are to be used. The Short Implants are characterized by 1.5mm supra-bony smooth collar, and 5.5mm infra-bony surface treated double threaded titanium.
  Interventions: Other: Single short implant

INTERVENTIONS:
Other: Double short implant — Patients receives 2 short implants to restore missing posterior teeth, loaded with splinted screw retained crowns.
  Arms: Two short implants
Other: Single short implant — Patients receives single short implants, loaded with single screw retained crowns.
  Arms: Single short implant

SUMMARY:
The aim of this study was to evaluate clinically and radiographically the splinted short implants' and single short implants' stability and bone condition before and after loading, in atrophic posterior mandibular alveolar ridges.

DETAILED DESCRIPTION:
A prospective study was conducted on 16 Patients with missing posterior molars. Group A: 8 patients had 2 short implants placed in atrophic posterior mandibular alveolar ridge. Group B: 8 patients had a single short implant placed in atrophic posterior mandibular alveolar ridge.

ELIGIBILITY:
Inclusion Criteria:

* Missing Posterior teeth, indicated for short implant placement.
* Residual alveolar ridge at 6-8 mm height and at least 7mm width.
* Healthy band of keratinized attached mucosa.
* Good Oral hygiene.
* Medically fit patient, free from relevant diseases.

Exclusion Criteria:

* Medically compromised patients.
* Imunnocompromised patients
* Patients with Para-functional habits.
* Smokers
* Poor Oral hygiene.
* Patient refuse to undergo the surgery.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Implant Stability | Immediately after the operation
  Implant stability was measured using Implant Stability Quotient (ISQ), a scale from 1 to 100. The ISQ scale has a non-linear correlation to micro-mobility. High stability means >70 ISQ, between 60-69 is medium stability and < 60 ISQ is considered as low stability.
Implant Stability | 3 months
  Implant stability was measured using Implant Stability Quotient (ISQ), a scale from 1 to 100. The ISQ scale has a non-linear correlation to micro-mobility. High stability means >70 ISQ, between 60-69 is medium stability and < 60 ISQ is considered as low stability.
Implant Stability | 6 months
  Implant stability was measured using Implant Stability Quotient (ISQ), a scale from 1 to 100. The ISQ scale has a non-linear correlation to micro-mobility. High stability means >70 ISQ, between 60-69 is medium stability and < 60 ISQ is considered as low stability.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Glantz PO, Nilner K. Biomechanical aspects of prosthetic implant-borne reconstructions. Periodontol 2000. 1998 Jun;17:119-24. doi: 10.1111/j.1600-0757.1998.tb00129.x. No abstract available. PMID 10337319
- [Background] Renouard F, Nisand D. Short implants in the severely resorbed maxilla: a 2-year retrospective clinical study. Clin Implant Dent Relat Res. 2005;7 Suppl 1:S104-10. doi: 10.1111/j.1708-8208.2005.tb00082.x. PMID 16137095
- [Background] Tallgren A. The reduction in face height of edentulous and partially edentulous subjects during long-term denture wear. A longitudinal roentgenographic cephalometric study. Acta Odontol Scand. 1966 Sep;24(2):195-239. doi: 10.3109/00016356609026127. No abstract available. PMID 5225747
- [Background] Nevins M, Al Hezaimi K, Schupbach P, Karimbux N, Kim DM. Vertical ridge augmentation using an equine bone and collagen block infused with recombinant human platelet-derived growth factor-BB: a randomized single-masked histologic study in non-human primates. J Periodontol. 2012 Jul;83(7):878-84. doi: 10.1902/jop.2012.110478. Epub 2012 Jan 5. PMID 22220770
- [Background] Chiapasco M, Casentini P, Zaniboni M. Bone augmentation procedures in implant dentistry. Int J Oral Maxillofac Implants. 2009;24 Suppl:237-59. PMID 19885448
- [Background] das Neves FD, Fones D, Bernardes SR, do Prado CJ, Neto AJ. Short implants--an analysis of longitudinal studies. Int J Oral Maxillofac Implants. 2006 Jan-Feb;21(1):86-93. PMID 16519186
- [Background] Neldam CA, Pinholt EM. State of the art of short dental implants: a systematic review of the literature. Clin Implant Dent Relat Res. 2012 Aug;14(4):622-32. doi: 10.1111/j.1708-8208.2010.00303.x. Epub 2010 Oct 26. PMID 20977606
- [Background] Thoma DS, Haas R, Tutak M, Garcia A, Schincaglia GP, Hammerle CH. Randomized controlled multicentre study comparing short dental implants (6 mm) versus longer dental implants (11-15 mm) in combination with sinus floor elevation procedures. Part 1: demographics and patient-reported outcomes at 1 year of loading. J Clin Periodontol. 2015 Jan;42(1):72-80. doi: 10.1111/jcpe.12323. Epub 2014 Dec 26. PMID 25418606
- [Background] Lemos CA, Ferro-Alves ML, Okamoto R, Mendonca MR, Pellizzer EP. Short dental implants versus standard dental implants placed in the posterior jaws: A systematic review and meta-analysis. J Dent. 2016 Apr;47:8-17. doi: 10.1016/j.jdent.2016.01.005. Epub 2016 Jan 19. PMID 26804969
- [Background] Misch CE, Steignga J, Barboza E, Misch-Dietsh F, Cianciola LJ, Kazor C. Short dental implants in posterior partial edentulism: a multicenter retrospective 6-year case series study. J Periodontol. 2006 Aug;77(8):1340-7. doi: 10.1902/jop.2006.050402. PMID 16937587
- [Background] Menchero-Cantalejo E, Barona-Dorado C, Cantero-Alvarez M, Fernandez-Caliz F, Martinez-Gonzalez JM. Meta-analysis on the survival of short implants. Med Oral Patol Oral Cir Bucal. 2011 Jul 1;16(4):e546-51. doi: 10.4317/medoral.16.e546. PMID 21196883
- [Background] Lum LB. A biomechanical rationale for the use of short implants. J Oral Implantol. 1991;17(2):126-31. PMID 1811063